CLINICAL TRIAL: NCT00935103
Title: The Effectiveness of Skill-Based HIV Psychoeducation in IV-Drug Abuser for Reducing High-risk Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 117
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Last update posted 2023-08-22 (Actual); Status verified 2009-07

CONDITIONS: Addiction; Risk Reduction Behaviour
Keywords: Addiction; Psychoeducation; Risk reduction behaviour; Drop in center (DIC)
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Psychoeducation (Active Comparator): Psycheducation
  Interventions: Behavioral: Psychoeducation
- Control (No Intervention): The control group will not take any intervention

INTERVENTIONS:
Behavioral: Psychoeducation
  Arms: Psychoeducation

SUMMARY:
The Effectiveness of Skill-Based HIV Psychoeducation in IV-Drug abuser for reducing high-risk behavior

ELIGIBILITY:
Inclusion Criteria:

Age more than 18 years old Dependency to opioid drugs (Positive result of Urin addiction test)

Exclusion Criteria:

suicide attempt not tendency for including to the study receiving treatment for addiction in recent months.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
IV usage of opioid | 12 months
  The number of usage by interview

SECONDARY OUTCOMES:
Usage of condom and safety syringe | 12 months
  the number of usage by interview